CLINICAL TRIAL: NCT03865368
Title: Immediate Effects of Whole Body Vibration on Hemodynamic Response and Fatigue in Normotensive Patients With Obesity
Brief Title: Immediate Effects of Whole Body Vibration on Hemodynamic Response and Fatigue in Normotensive People With Obesity
Acronym: RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Tülay Çevik, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Okan_University
Record Dates: First submitted 2019-02-27; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Obesity; Blood Pressure; Whole Body Vibration; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Active Whole Body Vibration (aWBVT) group, performed ten dynamic standard exercises on a vibration platform. The vibration protocol lasted for 15 minutes, in a frequency of 30 Hz and amplitude of 2 mm. Control group performed only ten dynamic standard exercises with no vibration application. Blood Pressure, heart rate, saturated oxygen were measured for the hemodynamic response. Modified Borg Dyspnoea Scale (MBDS) and The Borg Rating of Perceived Exertion (BRPE) Scale were used in order to evaluate fatigue level. All evaluations were performed at the beginning of the study, at the end of the session and at the recovery period
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Whole Body Vibration Training (Experimental): Exercises were taught during the first session, active training was done in the second session, and acute evaluations were made during the third session. Both groups performed the dynamic exercises, under supervision, on the whole body vibration device with 10-second rest intervals. Throughout the WBVT session, the vibration amplitude was set to 2 mm and exercise frequency 30 Hz.
  Interventions: Other: Whole Body Vibration Training
- Control Group (Active Comparator): The same exercises as the aWBVT group were performed on the vibration platform, with the vibration application turned off
  Interventions: Other: Whole Body Vibration Training

INTERVENTIONS:
Other: Whole Body Vibration Training — Whole Body Vibration Training (WBVT) method has been used as an alternative to conventional strengthening exercises. In this method, the patient stands on the platform of the WBVT device in a static position or performs dynamic exercises, the mechanical vibration produced by the device is transferred to the body
  Other Names: Standard Exercise

SUMMARY:
Whole Body Vibration Therapy (WBVT) has been identified as a useful tool to increase peripheral blood flow. The present study aimed at how dynamic exercises with WBVT immediate effect on hemodynamic response and fatigue parameters in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between age 18-65 with Body Mass Index (BMI) of >29.9 kg/m2

Exclusion Criteria:

* Unstable hypertensive patients
* History of cardiovascular, neurologic, or orthopedic diseases,
* Presence of knee prosthesis, hip replacement
* Chronic inflammatory disease,
* Anti-inflammatory treatment
* Cognitive impairments
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Heart rate | "20 minute"
  Heart rate was evaluated from the brachial artery using a sphygmanometer.
Blood pressure | "20 minute"
  Blood pressure was evaluated using a sphygmomanometer.

SECONDARY OUTCOMES:
Fatigue | "20 minute"
  Borg's Rating of Perceived Exertion Scale. Minimum score: 6 Maximum score: 20 The Borg Rating of Perceived Exertion scale helps estimate activity intensity.

OTHER OUTCOMES:
Change in Dyspnea | "20 minute"
  Modified Borg Dyspnea Scale Minimum score 0: breathing is causing no difficulty Maximum score 10: breathing difficulty is maximal

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Sports Laboratory, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided